CLINICAL TRIAL: NCT07061379
Title: Patient Reported Outcome Measurements (PROMs) Impact on Clinical Outcome in firsT Line settIng Non- Small-Cell Lung Cancer (NSCLC) According to Chemo- Immunotherapy reGimen (PROMOTING)
Brief Title: Patient Reported Outcome Measurements (PROMs) Impact on Clinical Outcome in firsT Line settIng Non- Small-Cell Lung Cancer (NSCLC) According to Chemo- Immunotherapy reGimen
Acronym: PROMOTING
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: AOU Città della Salute e della Scienza di Torino - Presidio Molinette (Unknown); Fondazione Policlinico Campus Bio-Medico (Unknown); ASST Lariana, Como (Unknown); IRCCS Istituto Nazionale dei Tumori (Unknown); ASST Grande Ospedale Metropolitano Niguarda (Other); IRCCS San Gerardo dei Tintori, Monza (Unknown); ASST Spedali Civili di Brescia (Unknown); Policlinico San Matteo Pavia (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Ospedale Vincenzo Monaldi (Unknown)
Responsible Party: Principal Investigator, Sara Oresti, MD, IRCCS San Raffaele
Other Study IDs: PROMOTING
Record Dates: First submitted 2025-06-20; First posted 2025-07-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: PROMs
Keywords: NSCLC; immunotherapy
MeSH Terms: interventions — Carboplatin; cemiplimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: patient treated with chemo-ICI regimen as first line therapy: Cohort A: Carboplatin/Cisplatin+Pemetrexed+Pembrolizumab/Cemiplimab (Keynote 189, EmpowerLung 3) for 4 cycles and then maintenance with Pemetrexed+Pembrolizumab/Cemiplimab up to 2 years or disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin/Cisplatin+Pemetrexed+Pembrolizumab/Cemiplimab for 4 cycles and then maintenance with Pemetrexed+Pembrolizumab/Cemiplimab up to 2 years or disease progression or unacceptable toxicity
- Cohort B: patient treated with double ICI-chemo regimen as first line therapy: Cohort B:
  Carboplatin/Cisplatin+Pemetrexed+Nivolumab+Ipilimumab (CheckMate9LA) for 2 cycles and then maintenance with Nivolumab q21 and Ipilimumab q42 up to 2 years or disease progression or unacceptable toxicity
  Interventions: Drug: Carboplatin/Cisplatin+Pemetrexed+Nivolumab+Ipilimumab for 2 cycles and then maintenance with Nivolumab q21 and Ipilimumab q42 up to 2 years or disease progression or unacceptable toxicity

INTERVENTIONS:
Drug: Carboplatin/Cisplatin+Pemetrexed+Pembrolizumab/Cemiplimab for 4 cycles and then maintenance with Pemetrexed+Pembrolizumab/Cemiplimab up to 2 years or disease progression or unacceptable toxicity — Cohort A: Carboplatin/Cisplatin+Pemetrexed+Pembrolizumab/Cemiplimab (Keynote 189, EmpowerLung 3) for 4 cycles and then maintenance with Pemetrexed+Pembrolizumab/Cemiplimab up to 2 years or disease progression or unacceptable toxicity
  Groups: Cohort A: patient treated with chemo-ICI regimen as first line therapy
Drug: Carboplatin/Cisplatin+Pemetrexed+Nivolumab+Ipilimumab for 2 cycles and then maintenance with Nivolumab q21 and Ipilimumab q42 up to 2 years or disease progression or unacceptable toxicity — Cohort B:
  Carboplatin/Cisplatin+Pemetrexed+Nivolumab+Ipilimumab (CheckMate9LA) for 2 cycles and then maintenance with Nivolumab q21 and Ipilimumab q42 up to 2 years or disease progression or unacceptable toxicity
  Groups: Cohort B: patient treated with double ICI-chemo regimen as first line therapy

SUMMARY:
A multicenter, national pharmacological observational study that has as its overall goal to implement a set of validated and agreed upon European-wide questionnaires (PROMs - patient's reported outcomes) to assess patients' perceptions of aspects of their lives based on the treatment they are receiving.

Specifically, with the research we present here, we aim to obtain data on patients' health and condition, including quality of life, symptom status, physical function, mental health (anxiety and depression), sleep quality, and sexuality as useful indicators not only of patient well-being but also of the effectiveness of the treatment itself.

The study involves the following: patients will be asked to complete online questionnaires at the following timepoints: before the start of treatment, after 4 and 8 treatment cycles, and at disease progression.

Data will also be collected regarding the patient's oncological medical history, treatment performed, response to treatment at CT/PET reevaluations, any toxicities that arose during treatment.

DETAILED DESCRIPTION:
Patient-reported outcomes measures (PROMs) are tools to assess patients' views on aspects of their health and condition, including health-related quality of life, symptom status, physical function and mental health. In medical oncology, PROMs are emerging as useful indicators not only of patient well-being, but also of treatment efficacy. Measurement of quality of life (QoL) has an intrinsic role in the definition of treatment value and, in the absence of head-to-head comparisons showing differences in overall survival or other traditional endpoints, comparison in terms of QoL can usefully inform the choice among alternative treatment options. The recent availability of alternative strategies in advanced NSCLC, in particular different combination therapies in first line setting, requires models to support clinical decision in tailoring individual treatments. In this model, the integration of PROMs could be essential in promoting a patient-centered approach to cancer care.

EORTC QLQ-C-30, exploring general functioning, and EORTC LC-13, specific for lung cancer are the most used PROMs tools in thoracic oncology.

QoL is a complex and composite outcome, which includes different aspects of patients' well-being, such as anxiety, depression and emotional stress. The latter has been measured in patients with lung cancer using PHQ-9 and Generalized Anxiety Disorder 7-item scales. Of note, a significant association with reduced response and worse survival upon immunotherapy was reported, suggesting an impact of emotional stress on patients' immune system and consequently on treatment outcomes.

Considering the broad effect of immunotherapy on the endocrine system and hormones' functions, it is likely that sexual health and sleep, other nuances of the QoL field, could be also affected by immunotherapy. So far, both sexual and sleep dysfunctions have been poorly explored in clinical trials. Furthermore, "time toxicity" defined as number of days with physical contact with healthcare system, could significantly affect patients' emotional distress sphere and has never been explored in NSCLC upon chemo-immunotherapy combinations.

Based on these assumptions, we believe that chemo-ICI (4 cycles of platinum-based doublet chemotherapy + anti- PD-1 followed by single agent chemo and immunotherapy maintenance) or double-ICI chemo (2 cycles of platinum-based doublet chemotherapy + anti-PD-1 and anti-CTLA-4, followed by maintenance with combo immunotherapy) regimens may have distinct effects on several QoL domains. This could be due to the intrinsic differences in the drugs used (i.e. addition of anti-CTLA-4 agents), treatment related toxicities and different tumor shrinkage activity.

The present study aims to compare QoL by validated questionnaires (EORTC QLQ-C-30, EORTC LC13) in the two above mentioned cohorts of patients with metastatic lung adenocarcinoma, having an additional focus in sexual (EORTC QLQ-SH-22), emotional stress (PHQ-9, Generalized Anxiety Disorder 7-item scale) and sleep disorders (PSQI) as previously reported. Time toxicity will be measured by analyzing the time patients spend in contact with healthcare system, such as visits and treatment. A defined cut off considers time toxicity severe when it exceeds 20% of the total care time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of Stage IV NSCLC with PD-L1 <50%, without actionable genomic alterations
* Signed Informed Consent Form (ICF) to the study
* Patients eligible to receive first line treatment with combo chemo-immuno treatments as standard of care

Exclusion Criteria:

- Patients unable to fill the questionnaires due to neurological comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of unresectable or advanced NSCLC eligible for first line chemo- ICI (Cohort A) or double ICI-chemo (Cohort B) regimens.
  Up to 50 patients with squamous histology, treated with any chemo- immunotherapy scheme will be monitored for QoL parameters as a prospective exploratory observational cohort and will not be included in the sample size calculation.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate what kind of first line treatment for metastatic lung adenocarcinoma has a better impact on quality of life of the patients | Baseline, after 4 cycles
  QoL domains assessed by EORTC QLQ-C-30 and LC13 at baseline and after 4 cycles. All questionnaires used in this study are validated questionnaires

SECONDARY OUTCOMES:
To assess the impact on overall survival of all the PROMs items under investigation | After 4 cycles, after 8 cycles, and at disease progression
  * QoL domains assessed by EORTC QLQ-C-30 and LC13 after 8 cycles of treatment and at disease progression
  * Sleep (PSQI), emotional stress (PHQ-9, GAD 7-item scale), sexual health ((EORTC QLQ-SH- 22) and time toxicity after 4 cycles, 8 cycles, and at disease progression
  * Overall Survival

OTHER OUTCOMES:
- To assess the impact on overall survival of all the PROMs items under investigation in squamous NSCLC | After 4 cycles, after 8 cycles and at disease progression
  QoL domains assessed by EORTC QLQ-C-30 and LC13 between double ICI-chemo or chemo- ICI regimens in patients with metastatic squamous NSCLC after 4 cycles, 8 cycles, and at disease progression.
- To assess the impact on PFS and RR in patients receiving different first line regimens | Baseline, after 4 cycles, after 8 cycles and at disease progression
  Progression-Free Survival (PFS) and Response Rate (RR) in each Cohort

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided